CLINICAL TRIAL: NCT04638127
Title: PREEMIE PROGRESS: A Family Management Program for Parents of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ashley Weber, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-0475; 1K23NR019081 (NIH)
Record Dates: First submitted 2020-10-22; First posted 2020-11-20 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Premature Infant Disease; Family Research; Parent-Child Relations; Self Efficacy; Patient Engagement; Patient Empowerment; Parenting; Chronic Conditions, Multiple
Keywords: neonatal intensive care unit; prematurity; family management; self-management; patient education
MeSH Terms: conditions — Patient Participation; Multiple Chronic Conditions; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREEMIE PROGRESS (Experimental): PREEMIE PROGRESS is an innovative, video-based intervention that applies evidence-based family management theories to better equip parents to meet the chronic, complex healthcare needs of their preterm infant.
  Interventions: Behavioral: PREEMIE PROGRESS
- Attention Control (Active Comparator): To maintain their attention, control parents will view "Welcome Videos" that explain hand hygiene, visitor IDs, parking, etc. on their mobile devices.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: PREEMIE PROGRESS — PREEMIE PROGRESS is a video-based training program for parents of preterm infants hospitalized in the neonatal intensive care unit (NICU).
  Arms: PREEMIE PROGRESS
Behavioral: Attention Control — usual care and welcome videos
  Arms: Attention Control

SUMMARY:
The purpose of this study is to refine and pilot test a mobile health (mHealth), video-based family management program for parents of preterm infants hospitalized in the Neonatal Intensive Care Unit (NICU). By moving beyond the basic infant care tasks taught by parenting programs and instead comprehensively training parents to use evidence-based family management skills, we hypothesize that our intervention, called PREEMIE PROGRESS, will better equip parents to meet the chronic, complex healthcare needs of their preterm infant.

DETAILED DESCRIPTION:
Increasing numbers of very preterm infants are surviving and have chronic, complex healthcare needs due to prematurity. These infants experience increased healthcare utilization, long durations of stay in the Neonatal Intensive Care Unit (NICU), and are at high risk of developing prematurity-related complications. As a result, their care is complex, and families need structured training to effectively understand, monitor, and manage their infant's care. PREEMIE PROGRESS is an innovative, video-based intervention that applies evidence-based family management theories to better equip parents to meet the chronic, complex healthcare needs of their preterm infant. This research aims to 1) refine a novel family management program, called PREEMIE PROGRESS, through iterative usability and acceptability testing and 2) test feasibility and acceptability of the refined intervention and study procedures in a pilot randomized controlled trial. This project will use implementation science tools and approaches to refine the intervention and study procedures to ensure that PREEMIE PROGRESS addresses key program elements that will be important for future adoption and implementation in NICU settings. We anticipate that the intervention will decrease parent anxiety and depression, increase infant weight gain and receipt of mother's milk, and reduce neonatal healthcare utilization. The long-term goal of this project is to develop, test, and translate into NICU practice an efficacious family management intervention for parents of preterm infants. Dr. Weber will significantly advance nursing science through this project by obtaining preliminary feasibility and acceptability data for a scalable and sustainable intervention to facilitate family management and improve parent-infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking parents
* Parents preterm infants born 25 0/7-31 6/7 weeks gestational age (GA)
* Parents who had a singleton or twin birth
* Parents 18 years of age or older

Exclusion Criteria:

* Mothers too ill (serious maternal complications, medications that impact alertness/ orientation) to provide informed consent
* Infants with imminent or probable death based on the healthcare team's judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley M Weber, PhD, RN, RNC-NIC, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Weber A, Bakas T, Oudat Q, Parikh NA, Lambert J, Tubbs-Cooley HL, Rice J, Voos K, Rota M, Kaplan HC. An Internet-Based and Mobile Family Management Intervention for Mothers of Very Preterm Infants Hospitalized in the Neonatal Intensive Care Unit (the Preemie Progress Program): Pilot Randomized Controlled Trial. JMIR Form Res. 2025 May 21;9:e66073. doi: 10.2196/66073. PMID 40397935

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PREEMIE PROGRESS | Attention Control
Started | 33 | 31
Completed | 16 | 26
Not Completed | 17 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREEMIE PROGRESS | Attention Control | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of mothers (in years)
  years | 29.1 (6.7) | 30.5 (4.3) | 29.8 (5.7)
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Infant gestation at birth (wks) | 29.2 (1.8) | 29.3 (2.1) | 29.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 17 | 23 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 29 | 59
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 10 | 23
  White | 18 | 17 | 35
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 31 | 64
Birth weight (g) [Mean (Standard Deviation); unit: grams] | 1253.9 (392.4) | 1286.2 (359.2) | 1269 (374)
Income (in $10,000) [Mean (Standard Deviation); unit: Annual income in $10,000] | 47000 (39000) | 44000 (39000) | 45400 (39000)
PROMIS (Patient-Reported Outcomes Measurement Information System)8a Anxiety [Mean (Standard Deviation); unit: T-score] — T-scores are reported. A PROMIS (Patient-Reported Outcomes Measurement Information System) T-score is a standardized score that helps compare an individual's score to the general population. The T-score is a score on a scale where 50 represents the average for the US general population. Each 10-point change represents one standard deviation (SD). A T-score of 75 or greater indicates clinically significant, severe symptoms. Higher T-scores indicate a higher level of the concept being measured. For example, a higher anxiety T-score would indicate more anxious symptoms.
  T-score | 53.4 (8.8) | 57.3 (76.9) | 55.2 (9.7)
PROMIS (Patient-Reported Outcomes Measurement Information System)8a Depression [Mean (Standard Deviation); unit: T-score] — T-scores are reported. A PROMIS (Patient-Reported Outcomes Measurement Information System) T-score is a standardized score that helps compare an individual's score to the general population. The T-score is a score on a scale where 50 represents the average for the US general population. Each 10-point change represents one standard deviation (SD). A T-score of 75 or greater indicates clinically significant, severe symptoms. Higher T-scores indicate a higher level of the concept being measured. For example, a higher depression T-score would indicate more depressive symptoms.
  T-score | 48.1 (8.6) | 49.3 (8) | 48.7 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Maternal Self-Rating of Depression
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) 8a Higher scores indicate higher levels of depression: T-score: standardized score mean of 50 and standard deviation (SD) of 10 The T-score is a score on a scale where 50 represents the average for the US general population (minimum of 8a Short Form is 38.2, maximum is 81.3). Each 10-point change represents one standard deviation (SD). A T-score of 75 or greater indicates clinically significant, severe symptoms.
Time Frame: Assessed at Baseline14 days post-baseline (T2), 28 days post-baseline (T3), and 30 days after infant discharge from the NICU (T4). Change from Baseline to 30 days after infant discharge from the NICU (T4) Reported.
Population: The percent of videos mothers watched were controlled in our analyses showing data trends as change scores. At each follow-up time point [14 days post-baseline (T2), 28 days post-baseline (T3), and 30 days after infant discharge from the NICU (T4)], we computed mean differences and 95% CI between groups to evaluate trends in outcomes. Reported here are mean (SE) in change scores from Baseline to 30 days after infant discharge from the NICU (T4).
Measure: Mean (Standard Error); unit: T-score mean changes
Arm/Group | PREEMIE PROGRESS | Attention Control
Number analyzed (Participants) | 33 | 31
T-score mean changes
  T2 - Baseline | -3.75 (1.70) | -4.08 (1.42)
  T3 - Baseline | -2.21 (1.58) | -2.50 (1.35)
  T4 - Baseline | -4.08 (1.42) | -3.75 (1.70)

2. Primary Outcome: Maternal Self-Rating of Anxiety
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) 8a Higher scores indicate higher levels of anxiety: T-score: standardized score mean of 50 and standard deviation (SD) of 10 The T-score is a score on a scale where 50 represents the average for the US general population (minimum of 8a Short Form is 38.2, maximum is 81.3). Each 10-point change represents one standard deviation (SD). A T-score of 75 or greater indicates clinically significant, severe symptoms.
Time Frame: Assessed at Baseline, 14 days post-baseline (T2), 28 days post-baseline (T3), and 30 days after infant discharge from the NICU (T4). Change from Baseline to 30 days after infant discharge from the NICU (T4) Reported.
Population: The percent of videos mothers watched were controlled in our analyses showing data trends as change scores. At each follow-up time point [14 days post-baseline (T2), 28 days post-baseline (T3), and 30 days after infant discharge from the NICU (T4)], we computed mean differences and 95% CI between groups to evaluate trends in outcomes. Reported here are mean (SE) in change scores from Baseline at each time point in the study.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | PREEMIE PROGRESS | Attention Control
Number analyzed (Participants) | 33 | 31
T-score
  T2-Baseline | -3.08 (1.74) | -1.96 (1.52)
  T3-Baseline | 2.87 (1.77) | -3.91 (1.53)
  T4-Baseline | -4.67 (1.59) | -7.54 (1.93)

3. Primary Outcome: Receipt of Exclusive Mother's Human Milk
Description: Number of infants receiving exclusive mother's milk were recorded and percent of infants was calculated from the total number number of infants receiving enteral feeds. Infants were marked as receiving exclusive mother's milk if all feeds were mother's milk (i.e., infant did not receive donor milk or formula).
  Percent of infants receiving exclusive mother's milk = Number of infants receiving exclusive mother's milk / Number of infants on enteral feeds
Time Frame: Assessed at Baseline, 14 days post-baseline (T2), 28 days post-baseline (T3).
Population: Assessed at Baseline, 14 days post-baseline (T2), 28 days post-baseline (T3).
Measure: Count of Participants; unit: Participants
Arm/Group | PREEMIE PROGRESS | Attention Control
Number analyzed (Participants) | 33 | 30
Participants
  Baseline | 17 | 18
  T2: number analyzed (Participants) | 31 | 29
  T2 | 13 | 15
  T3: number analyzed (Participants) | 26 | 28
  T3 | 14 | 10

4. Primary Outcome: Change in Fenton 2013 Growth Calculator Z-scores From Birth to 36 Weeks Corrected Gestational Age
Description: Change in Z score weight from birth to 36 weeks corrected gestational age (or at discharge if earlier) was calculated using PediTools Fenton 2013 Growth Calculator for Preterm Infants. Z-scores are the number of standard deviations above or below a growth chart's center (mean) curve. A Fenton preterm growth chart Z-score of 0 means the infant's growth measurement (e.g., weight) is at the average (mean) for their age and sex. Changes in Z-scores tell if a second measurement is closer or further away from the growth chart center than the previous measurement. Change in Z-score of 0 means the infant's percentile on the growth chart did not change. Higher Z scores indicate increased growth acceleration. The Academy of Nutrition and Dietetics considers Z score changes less than -0.8 to indicate growth failure. Normal growth during NICU hospitalization is defined as a z-score change of -0.79 to 0.79.
  Z score Δ = [Zscore at 36 weeks corrected gestational age] - [Zscore at birth]
Time Frame: Z scores were calculated at 36 weeks corrected gestational age (or at discharge if earlier) and at birth.
Population: Z score Δ = [Zscore at 36 weeks corrected gestational age] - [Zscore at birth]
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | PREEMIE PROGRESS | Attention Control
Number analyzed (Participants) | 33 | 31
Z-score | -0.8 [-1.36 to -0.51] | -0.72 [-1.11 to -0.39]

5. Primary Outcome: NICU Length of Stay
Description: Days of NICU hospitalization (calculated from days between date of birth to date of discharge from NICU)
Time Frame: Date of NICU discharge will be assessed until study completion, with maximum of 1 year
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Attention Control | PREEMIE PROGRESS
Number analyzed (Participants) | 31 | 33
days | 68.3 (36.3) | 57.2 (23.4)

6. Primary Outcome: Infant Hospital Readmissions and Emergency Department Visits Within 30 Days of Infant Discharge - YES Response
Description: The infant's electronic health record was reviewed for hospital readmissions and emergency department visits within 30 days of infant discharge. Mothers were also asked "Did your infant have any re-hospitalizations or emergency department visits within 30 days of discharge?", to ensure all rehospitalizations and ED visits were captured.
Time Frame: Thirty days after infant discharge from the NICU.
Population: Coded as Yes/No and extracted from the infant's electronic health record. Mothers were also asked "Did your infant have any re-hospitalizations or emergency department visits within 30 days of discharge?", to ensure all rehospitalizations and ED visits were captured.
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control | PREEMIE PROGRESS
Number analyzed (Participants) | 31 | 33
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: Assessed at Baseline, 14 days post-baseline (T2), 28 days post-baseline (T3), and 30 days after infant discharge from the NICU (T4).
Arm/Group | Attention Control | PREEMIE PROGRESS
All-Cause Mortality (participants affected / at risk) | 0/31 | 1/34
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/34
Other Adverse Events (participants affected / at risk) | 3/31 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attention Control (N=31) | PREEMIE PROGRESS (N=34)
Psychological Distress, Clinical significant Anxiety or Depression (Psychiatric disorders) | 3 (3) | 0 (0) — self-reported psychological distress or clinically significant symptoms of anxiety or depression (i.e., T-Score >75.0 on PROMIS8a Anxiety or PROMIS8a Depression)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT04638127/Prot_SAP_000.pdf